CLINICAL TRIAL: NCT00269958
Title: A Double-Blind, Phase II, Placebo-Controlled Study to Determine the Safety and Efficacy of r-HuEPO in Reducing Transfusion Requirements in Patients Undergoing Total Hip Joint Replacement Surgery
Brief Title: A Study to Evaluate the Safety and Efficacy of Epoetin Alfa Versus Placebo to Reduce the Need for Blood Transfusions and Reduce the Occurrence of Severe Anemia During the Time Period Surrounding Total Hip Replacement Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen-Ortho Inc., Canada (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR005887
Record Dates: First submitted 2005-12-22; First posted 2005-12-26 (Estimated); Last update posted 2011-05-17 (Estimated); Status verified 2010-04

CONDITIONS: Anemia
Keywords: hip replacement; hip replacement surgery; surgery; anemia; transfusions; blood transfusions
MeSH Terms: conditions — Anemia | interventions — Epoetin Alfa

INTERVENTIONS:
Drug: epoetin alfa

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of two different dosing schedules of epoetin alfa versus placebo for decreasing the need for blood transfusions and preventing the occurrence of severe anemia during the period of time around total hip replacement surgery. Epoetin alfa is a genetically engineered protein that stimulates red blood cell production.

DETAILED DESCRIPTION:
Major surgical procedures may require blood transfusions both during and after the operation. Agents that can increase the rate of red blood cell production would reduce the need for blood transfusions and reduce the occurrence of anemia. Epoetin alfa is a genetically engineered form of a natural hormone, erythropoietin, that is used to treat anemia by stimulating red blood cell production. This is a randomized, double-blind, placebo-controlled, parallel group, multicenter study in patients scheduled for total hip replacement surgery. This study will assess the effectiveness of epoetin alfa (starting either 5 or 10 days before hip replacement surgery and continuing though 3 days after surgery) in reducing the need for blood transfusions and the occurrence of anemia during the time period surrounding surgery. Hip replacement can be either the initial implant surgery or a second surgery on the same hip. Eligible patients will be assigned to one of three treatment groups. Group 1 will receive daily placebo injections under the skin for 14 days; Group 2 will receive a longer (14-day) course of daily epoetin alfa injections under the skin; and Group 3 will receive a shorter (9-day) course of daily epoetin alfa injections under the skin. Patients in Groups 2 and 3 will receive 300 units of epoetin alfa per kilogram of body weight per day in each daily injection. All patients will receive oral iron supplementation beginning 3 weeks prior to surgery and continuing through 1 week after surgery. All patients will also receive low-dose coumadin (sodium warfarin) for 7 days after surgery to prevent clotting in the deep veins. Effectiveness will be determined by the number of patients requiring transfusions and the number of patients who develop anemia (as measured by a hemoglobin level < 80 grams per liter). Effectiveness will also be determined by the total number of transfusions required, changes in red blood cell variables (hemoglobin, hematocrit, the number of developing red blood cells (reticulocytes), changes in the iron stores in the patient's blood, intensity of nursing care required, well-being assessments (measures of pain, shortness of breath, and energy level), and the number of days in the hospital after surgery. Safety evaluations will include the incidence of blood clots in the deep veins of the lower limbs, the incidence and severity of other adverse events, and changes in clinical laboratory test results and vital signs. The study hypothesis is that patients treated with epoetin alfa before, during, and after hip replacement surgery will require fewer blood transfusions and have a reduced occurrence of anemia compared with patients treated with placebo, and that the shorter course of epoetin alfa dosing (9 days) is as effective as the longer epoetin alfa course (14 days). 300 units epoetin alfa per kilogram (U/kg) injected under the skin 5 or 10 days before surgery, the day of surgery, and 3 days after surgery; or placebo injection for 14 days. Subjects receiving epoetin alfa for 5 days also received placebo for 5 days before starting epoetin alfa.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective, first-time hip-replacement surgery or a second hip-replacement surgery (with surgery taking place within 48 hours of the scheduled time)
* having a baseline hemoglobin between 110 and 160 grams per liter
* with no significantly abnormal values for laboratory tests that would indicate an impaired ability to respond to epoetin alfa.

Exclusion Criteria:

* Patients with a primary hematologic disease
* having any clinically significant disease/dysfunction of the neurologic, pulmonary, endocrine, cardiovascular, gastrointestinal, or genitourinary systems
* who have had a seizure disorder in the past 5 years, or who are currently on anticonvulsant therapy
* having uncontrolled high blood pressure
* currently experiencing an ongoing blood loss

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Study Completion 1991-12 (Actual)

PRIMARY OUTCOMES:
Proportion of patients needing blood transfusions; proportion of patients who develop anemia (defined as hemoglobin <80 grams per liter).

SECONDARY OUTCOMES:
Number of blood units transfused; changes in red cell variables (hemoglobin, hematocrit, and reticulocyte counts); iron stores; nursing needs; scores on well-being tests; number days in hospital after surgery; deep vein clots and other adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Ortho Inc. Clinical Trial, Study Director — Janssen-Ortho Inc., Canada

REFERENCES:
- See also: A study to evaluate the efficay of epoetin alfa to reduce the need for blood transfusions and reduce the occurrence of severe anemia during the time period surrounding total hip replacement surgery — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=363&filename=CR005887_CSR.pdf